CLINICAL TRIAL: NCT07244900
Title: Effects Of Conventional Physical Therapy With And Without Action Observation Therapy On Freezing Of Gait And Functional Mobility In Participants With Parkinson's Disease: A Randomised Clinical Trial
Brief Title: Conventional Physical Therapy Action Observation Therapy on Freezing of Gait and Functional Mobility in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kiran Maqsood
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease; Neuro-Degenerative Disease
Keywords: Parkinson's Disease; Balance; Freezing of Gait; Mobility; Function
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This study follows a parallel group design, involving two groups: a control group and an experimental group. Participants in both groups will receive treatment concurrently but under different conditions. The control group will receive the standard or conventional intervention, while the experimental group will receive the modified or additional treatment being investigated. Comparisons between the groups will be made to evaluate the effectiveness of the experimental intervention.
Who Masked: Outcomes Assessor
Masking Description: This study will use a single-blind masking design, in which the outcome assessor will be blinded to group allocation. Participants and therapists will be aware of the intervention assigned, but the assessor responsible for data collection and analysis will not have access to group assignment information to minimize assessment bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy Group (Active Comparator): This group included conventional physical therapy that contains isometric exercise, stretching techniques, and strength and balance training.
  Interventions: Other: Conventional Physical Therapy
- Experimental Group (Experimental): This group included action observation therapy in addition to conventional physical therapy, in which small videos containing specific task will be made available to follow to the participants.
  Interventions: Other: Action Observation plus conventional Physical Therapy

INTERVENTIONS:
Other: Conventional Physical Therapy — Group A received conventional physical therapy treatment. The CPT program consists of isometric exercises, stretching, and strength training based on the patient's physical condition and the severity of functional mobility and freezing of Gait.
  Arms: Conventional Physiotherapy Group
Other: Action Observation plus conventional Physical Therapy — Group B was given action observation therapy with conventional physical therapy treatment. In AOT, the therapist showed small video clips of different goal-directed tasks to participants, and they were asked to follow every step and movement. The therapist maintained the patient's attention with verbal feedback
  Arms: Experimental Group

SUMMARY:
The goal of this study is to determine the effects of action observation therapy with conventional physical therapy on freezing gait and functional limitation in participants with Parkinson's disease.

DETAILED DESCRIPTION:
Parkinson's disease is a neurodegenerative disorder that is characterized by rigidity, tremors, and bradykinesia, along with non-motor dysfunction. The exercise rehabilitation has a positive impact on motor and non-motor functions in individuals with Parkinson's disease. Conventional physical therapy (CPT) that involves isometric exercises, stretching techniques, and strength and balance training is useful to improve the severity of functional mobility and freezing of gait. In action observation therapy (AOT), small video clips of different goal-directed tasks were added to rehabilitation to determine the combined effects on outcome.

ELIGIBILITY:
Inclusion Criteria: The participants were included based on the UK Parkinson's Disease Society Brain Bank diagnostic criteria, with clinical findings supporting the diagnosis. The eligible participants were aged between 50 and 80 years, of both genders, labelled as stage ≤ 3, with a minimum of 2 years since being diagnosed with PD and a freezing of gait score of 9 or higher on FOG-Q, and able to understand and follow commands.

Exclusion Criteria:

The exclusion criteria were systemic disease and neurological issues that could affect the assessment and outcomes of treatment, implantation for deep brain stimulation, and visual or acoustic limitations.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in functional mobility | The assessment was made at baseline before the treatment session, and any change in mobility status was observed at the end of 6th week and 12th week after the intervention.
  The TUG is an efficient test that measures mobility and balance, requiring participants to rise from a chair, walk 3 meters, turn, walk back, and sit down. The time taken to complete this sequence is recorded, with longer times indicating potential mobility issues. A score of more than or equal to fourteen seconds indicates a high risk of falls.
Change in Freezing of gait | The freezing of gait was assessed at baseline, and any change in it was measured at the end of 6th week and 12th week after the intervention.
  The FOG-Q is a reliable tool for evaluating the effectiveness of treatment intervention on FOG for Parkinson's disease. The questionnaire consists of 6 items designed to assess the severity of freezing of gait. Each item is rated on a five-point Likert scale, with '0' indicating no symptoms and '4' indicating the most severe symptoms. The total score can range from 0 to 24, with higher scores indicating greater severity of freezing of gait.

CONTACTS AND LOCATIONS:
Overall Officials: Ishfaq Ahmed, PhD Physiotherapy, Study Director — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the study will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Three years after the publication of result findings
Access Criteria: Access to the de-identified individual participant data (IPD) and supporting documents will be available to qualified researchers affiliated with recognized academic or research institutions. Interested researchers may request access by submitting a written proposal outlining the study objectives and analysis plan to the principal investigator or corresponding author.
  Upon approval, the data (including de-identified participant-level datasets, study protocol, and statistical analysis plan) will be shared via a secure institutional data repository or encrypted email. Data will be provided solely for non-commercial, academic research purposes and must comply with applicable ethical and data protection standards.
URL: https://oric.uol.edu.pk/